CLINICAL TRIAL: NCT04067479
Title: Can Amino Acid Supplementation Augment the Anabolic Response in Tendon After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Chad C. Carroll, Assistant Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1704019133
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Tendinopathy
Keywords: tendon; amino acid; exercise
MeSH Terms: conditions — Tendinopathy; Motor Activity | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young (Experimental): 21-30 year old men and women Inclusion/Exclusion Criteria
  1. All subjects will be sedentary or recreationally active (sedentary: one day or less per week of aerobic or resistance exercise for at least a year or recreationally active: not training for competitive events).
  2. Age: 21-30 years
  3. Body mass index <35 kg•m-2,
  4. Chronic users of medications such as acetaminophen, ibuprofen, or prescription cyclooxygenase inhibitors will be excluded as these medications have been shown to alter tendon physiology.
  5. Individuals with diabetes will be excluded. Diabetes is thought to change the structure of tendon.
  6. Individuals with a history of tendon pain will be excluded, as chronic tendon pain is associated with changes in the structure of tendon.
  7. Persons with allergies/sentivitiy to amino acids or ingedianet of Cystal Light will be excluded.
  Interventions: Dietary Supplement: Amino Acids
- Older Adults (Experimental): Inclusion/Exclusion Criteria
  1. All subjects will be sedentary or recreationally active (sedentary: one day or less per week of aerobic or resistance exercise for at least a year or recreationally active: not training for competitive events).
  2. Age: 60-75 years
  3. Body mass index <35 kg•m-2
  4. Chronic users of medications such as acetaminophen, ibuprofen, or prescription cyclooxygenase inhibitors will be excluded as these medications have been shown to alter tendon physiology.
  5. Individuals with diabetes will be excluded. Diabetes is thought to change the structure of tendon.
  6. Individuals with a history of tendon pain will be excluded, as chronic tendon pain is associated with changes in the structure of tendon.
  7. Persons with allergies/sentivitiy to amino acids or ingedianet of Cystal Light will be excluded.
  Interventions: Dietary Supplement: Amino Acids

INTERVENTIONS:
Dietary Supplement: Amino Acids — Oral bolus of essential amino acids

SUMMARY:
The goal of this study is to determine if an oral provision of amino acids will enhance exercise-induced increases in markers of Achilles tendon collagen production.

DETAILED DESCRIPTION:
Tendon pain is a common complaint in older adults. The mechanisms contributing to the large number of tendon problems in older adults are not known. It has been shown that tendon cross-sectional area (CSA) is reduced with aging concurrent with a significant loss of tendon collagen. Exercise is used to reverse the loss of muscle mass with aging but surprisingly exercise interventions designed to reduce tendon problems in older people are relatively unexplored. In young adults, exercise stimulates tendon collagen synthesis and enhances the production of growth factors, which stimulate tendon collagen production. It is presumed that exercise-induced increase in collagen synthesis contributes to the increase in tendon stiffness and CSA noted in young adults after chronic resistance exercise (RE). In contrast, our preliminary work indicates that RE is not effective at reducing the effects of aging on tendon. The investigators have demonstrated that 12-weeks of RE does not lead to increases in tendon CSA or stiffness, even when skeletal muscle mass and strength are greatly enhanced. To prevent tendon injury, greater tendon CSA and stiffness aid in withstanding the force generated by trained skeletal muscle. Greater CSA and stiffness also optimize force transfer through tendon to maximize musculoskeletal function. Our findings indicate that RE is not an optimal intervention for reversing age-related changes in tendon properties. Novel interventions are clearly needed that will enhance collagen synthesis leading to an increase in tendon stiffness and CSA while also improving skeletal muscle mass and strength in older individuals. This study will evaluate the effectiveness of various methods for stimulating tendon collagen synthesis during a bout of acute exercise. Specifically, the investigators propose two approaches to this problem.

1. An acute bout of cycling exercise will enhance the release of growth factors leading to a larger increase in tendon collagen synthesis.
2. A bolus of amino acids given orally will increase the release of key stimulators of tendon collagen synthesis leading to enhanced collagen synthesis after acute exercise.

ELIGIBILITY:
Inclusion Criteria:

* 21-35 years or 60-80 years old

Exclusion Criteria:

* diabetes
* BMI>35
* acute illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, metabolic disorders, arthritis, or a history of neuromuscular problems.
* chronic pain medication users
* alcoholism
* competitive athletes
* pregnant women will be excluded
* Individuals with specific allergies to amino acids

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Achilles peritendinous concentrations of pro-collagen | 0-6 hours post consumption
  Peritendinous samples will be collected using microdialysis. Pro-collagen will be assessed using enzyme immunoassay kits
Amino Acid Levels | 0-6 hours post consumption
  Achilles peritendinous amino acid concentrations will be assess using high performance liquid chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Chad C Carroll, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No